CLINICAL TRIAL: NCT00493519
Title: Cephalic Phase in Anorexia Nervosa,Bulimia Nervosa and Obese Binge Eaters
Acronym: Cephalic 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TASMC-07-NV-219-CTIL
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-04

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
Keywords: Cephalic phase; Anorexia nervosa; Bulimia nervosa; obese binge eaters; VAS; EDI; shame-feed procedure
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: chocolate cake

SUMMARY:
The objective of this trial is to examine the cephalic phase insulin response (CPIR) and pancreatic polypeptide (PP) release as indicators of the cephalic phase occurrence and magnitude to palatable food stimulus in anorectic and bulimic subgroups as compared to healthy controls

DETAILED DESCRIPTION:
Food stimulation of gastric and pancreatic secretion is classically divided into cephalic, gastric and intestinal phases.

Cephalic phase refers to a simultaneous activation of gastrointestinal motility, gastric acid and pancreatic enzyme secretion ,as well as, release of hormones from the endocrine pancreas which occurs through activation of vagal -efferents as a result of food-related sensory stimuli such as taste and smell prior to nutrient absorption and which coincides with a thermogenic response.

Of the cephalic phase secretions, cephalic phase insulin release (CPIR) has received the most attention, but pancreatic polypeptide (PP) and glucagon responses have also been studied. While the magnitude of cephalic phase insulin release is relatively small (25% above baseline), pancreatic polypeptide increases 100% above baseline. The large magnitude of the PP response makes it a sensitive indicator of vagal activation to food stimuli.

In most experiments, subjects are either exposed to visual and olfactory stimulation by seeing and smelling the food stimulus or are required to perform a modified sham-feed, i.e. to taste, chew and then expectorate the food stimulus.

In general, cephalic phase are thought to be preparatory response before ingestion of food. Because of their small magnitude, the physiological significance of the cephalic phase hormonal responses has been largely discounted. However, there is evidence that experimental prevention of CPIR lead to hyperinsulinemia and hyperglycemia. Therefore, CPIR may contribute to glucose homeostasis /regulation. Moreover CPIR may be an indicator of hunger and could be important for understanding eating disorders.

In parallel with these hormonal secretion ,an increase in energy expenditure has also been observed . This thermogenic response to food is even greater with sham feeding than with normal feeding and is paralleled by changes in RQ showing enhanced carbohydrate oxidation.

Studies conducted in obese humans demonstrate exaggerated absolute magnitude of CPIR .However basal hyper-insulinemia which is typically observed in obese individuals may clouds this observation. Moreover, it has been hypothesized that CPIR is attenuated in obese when is expressed as a percentage of baseline and therefore they may not secrete enough insulin during pre-absorptive period to regulate postprandial glucose levels.

There is also evidence that obese people with insulin resistance have a reduced thermogenic response to feeding .

Only limited numbers of studies have been done on the cephalic phase in anorexia and bulimia. There are findings of a significant CPIR in anorexics as compared to controls which tends to rule out a deficient cephalic insulin response as a contributor to the self-starvation observed in anorexia nervosa. As to bulimics who often show endocrine abnormalities, their CPIR was only slightly differ or from controls.

These findings suggest more complex determinants of eating disorders than physiological state alone.

ELIGIBILITY:
Inclusion Criteria:

75 patients will be divided into the following 4 subgroups;

1. . 15 patients with anorexia nervosa.
2. . 15 patients with bulimia nervosa (purging type).
3. . 15 patients with binge eating disorder and obesity.
4. . 15 obese patients without eating disorder
5. . 15 Non-eating disordered normal weight patients.

Non diabetic and non-pregnant patients above 18 years of age without gastrointestinal diseases and without medications which can affect gastrointestinal motility and appetite.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-07; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
VAS, EDI, Blood test for glucose, insulin, PP, shame feed procedure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof., Principal Investigator — TASMC Israel
Locations (1):
- TASMC, Tel Aviv, Israel